CLINICAL TRIAL: NCT01366417
Title: Test for Preinjection Skin Preparation
Brief Title: Topical Antimicrobial Effectiveness Testing
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: C. R. Bard (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Other
Other Study IDs: 371.1.04.19.11
Record Dates: First submitted 2011-06-02; First posted 2011-06-06 (Estimated); Results first posted 2012-08-31 (Estimated); Last update posted 2025-12-11 (Actual); Status verified 2025-11

CONDITIONS: Antimicrobial Effectiveness
MeSH Terms: interventions — 2-Propanol

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: ChloraPrep One-Step — 1.5 ml applicator patient preoperative skin preparation
Drug: 70% isopropyl alcohol — Curity Alcohol Prep Pads
  Other Names: Positive Control

SUMMARY:
The primary objective of this study is to measure the antimicrobial effectiveness of ChloraPrep One-Step Frepp Applicator.

ELIGIBILITY:
Inclusion Criteria:

* in good general health
* have skin within 6 inches of the test sites that is free of tattoos, dermatoses, abrasions, cuts, lesions or other skin disorders.

Exclusion Criteria:

- topical or systemic antimicrobial exposure within 14 days prior to the Screen Visit

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2011-05; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad H Bashir, MD, Principal Investigator — Microbiotest
Locations (1):
- Microbiotest, Sterling, Virginia, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First subject/first visit: May 12, 2011 Last subject/last visit: June 8, 2011
Pre-assignment Details: 43 subjects entered screening phase.25 subjects had qualifying treatment day baseline counts and completed the study.
Groups:
- ChloraPrep One Step and 70% Isopropyl Alcohol: All subjects received a single topical treatment with both the test article (ChloraPrep One Step) and the positive control (Isopropyl Alcohol)
Period: Overall Study
Arm/Group | ChloraPrep One Step and 70% Isopropyl Alcohol
Started | 43
Signed Informed Consent | 43 (Microbial samples were taken from 43 subjects for screening baseline.)
Completed Screen Visit | 33 (33 subjects had qualifying screening bacterial counts and were eligible for the Treatment Visit)
Completed Treatment Visit | 28 (28 subjects were treated with ChloraPrep and 70% Isopropyl Alcohol (single topical treatment))
Completed the Study | 28 (treatment baseline microbial counts not available until after treatment; subjects not evaluable)
Discontinued Prior to Treatment | 5 (5 eligible subjects were not treated because enrollment target of 25 was met and enrollment closed.)
Excluded From Analysis | 3 (3 subjects did not have qualifying Treatment Day microbial counts and were excluded from analysis)
Completed | 25 (25 subjects included in the analysis)
Not Completed | 18

BASELINE CHARACTERISTICS:
Arm/Group | ChloraPrep One Step and 70% Isopropyl Alcohol
Number analyzed (Participants) | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 28
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 36 (16.71105)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 12
Region of Enrollment [Number; unit: participants]
  United States | 28

OUTCOME MEASURES:

1. Primary Outcome: Antimicrobial Efficacy
Description: Antimicrobial efficacy will be measured by the change (+/-) in bacterial count on the skin 30 seconds after a single application of test material relative to the baseline bacterial count.
Time Frame: 30 seconds after treatment
Population: subjects whose treatment day baseline microbial count met the qualification criteria and completed all assessments.
Measure: Mean (95% Confidence Interval); unit: log 10 colony forming units / cm^2
Groups:
- ChloraPrep One Step: All subjects received a single topical application of ChloraPrep One Step.
- 70% Isopropyl Alcohol: All subjects received a single topical application of 70% Isopropyl Alcohol.
Arm/Group | ChloraPrep One Step | 70% Isopropyl Alcohol
Number analyzed (Participants) | 25 | 25
log 10 colony forming units / cm^2 | 2.21 (0.1332) [1.95 to 2.48] | 2.25 (0.1332) [1.99 to 2.51]
Statistical Analysis 1: Comparison: ChloraPrep One Step; Hypothesis: ChloraPrep will meet or exceed the 1.0 log reduction in colony forming units/cm^2 at 30 seconds after application; Test type: Superiority or Other; p < 0.05, ANOVA; Mean Difference (Net) = 2.21, 95% CI 2-sided [1.95 to 2.48], Standard Error of Mean 0.133
Statistical Analysis 2: Comparison: 70% Isopropyl Alcohol; hypothesis: 70% Isopropyl Alcohol will meet or exceed 1.0 log 10 colony forming units / cm^2 at 30 seconds after treatment; Test type: Superiority or Other; p < 0.05, ANOVA; Mean Difference (Net) = 2.25, 95% CI 2-sided [1.99 to 2.51], Standard Deviation 0.133

2. Primary Outcome: Antimicrobial Efficacy
Description: Antimicrobial efficacy will be measured by the change (+/-) in bacterial count on the skin 10 minutes after a single application of test material relative to the baseline bacterial count.
Time Frame: 10 minutes after treatment
Population: Subjects whose Treatment Day Baseline bacterial counts met qualification criteria
Measure: Mean (95% Confidence Interval); unit: log 10 colony forming units / cm^2
Arm/Group | ChloraPrep One Step | 70% Isopropyl Alcohol
Number analyzed (Participants) | 25 | 25
log 10 colony forming units / cm^2 | 2.65 [2.39 to 2.92] | 2.60 [2.33 to 2.86]
Statistical Analysis 1: Comparison: ChloraPrep One Step; Hypothesis: ChloraPrep One Step will meet or exceed 2.0 log 10 reduction at 10 minutes after treatment; Test type: Superiority or Other; p < 0.05, ANOVA; Mean Difference (Net) = 2.65, 95% CI 2-sided [2.39 to 2.91], Standard Deviation 0.133
Statistical Analysis 2: Comparison: 70% Isopropyl Alcohol; Hypothesis: 70% Isopropyl Alcohol will meet or exceed 2.0 log 10 reduction at 10 minutes after treatment; Test type: Superiority or Other; p < 0.05, ANOVA; Mean Difference (Net) = 2.60, 95% CI 2-sided [2.33 to 2.86], Standard Deviation 0.133

ADVERSE EVENTS:
Arm/Group | ChloraPrep One Step and 70% Isopropyl Alcohol
Serious Adverse Events (participants affected / at risk) | 0/28
Other Adverse Events (participants affected / at risk) | 0/28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No